CLINICAL TRIAL: NCT01221948
Title: VANTAGE STUDY Vercise™ Implantable Stimulator for Treating Parkinson's Disease
Brief Title: Vercise Implantable Stimulator for Treating Parkinson's Disease
Acronym: VANTAGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5001
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Deep Brain Stimulation; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Boston Scientific Vercise Deep Brain Stimulation system will be implanted and each patient will serve as its own control.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): Rechargeable Deep Brain Stimulation System
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Rechargeable Deep Brain Stimulation System

SUMMARY:
The purpose of this study is to document patient outcomes, including effectiveness, safety, and health economic data, for the Boston Scientific implantable deep brain stimulation (DBS) Vercise™ system for bilateral stimulation of the subthalamic nucleus (STN) in the treatment of moderate to severe idiopathic Parkinson's Disease (PD).

DETAILED DESCRIPTION:
This is a multi-center, prospective, open label, non-randomized study which will use a within-patient control (each patient serves as his/her own control) to document patient outcomes, including effectiveness, safety, and health economic data for the Boston Scientific implantable deep brain stimulation (DBS) Vercise™ system for bilateral stimulation of the subthalamic nucleus (STN) in the treatment of moderate to severe idiopathic Parkinson's Disease (PD).

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of bilateral idiopathic PD with the presence of at least 2 of the following: resting tremor, rigidity, or bradykinesia.
2. Duration of bilateral idiopathic PD of more than five years.
3. Stable medications
4. UPDRS subset III score of ≥30 without medication.
5. Lack of dementia or depression.
6. Must improve with antiparkinsonian medication, but have some motor complications that are not well controlled by medications.
7. Must be an appropriate candidate for the surgical procedures required for bilateral STN DBS.
8. Is willing and able to comply with all visits and study related procedures
9. Patient understands the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed.

Key Exclusion Criteria:

1. Any intracranial abnormality or medical condition that would contraindicate DBS surgery.
2. Any finding in neuropsychological screening assessments that would contraindicate DBS surgery, including dementia.
3. Any significant psychiatric problems, including unrelated clinically significant depression.
4. Any current drug or alcohol abuse.
5. Any history of recurrent or unprovoked seizures.
6. Frequent falls while receiving good medication therapy without dyskinesias (on-state).
7. Any prior movement disorder treatments that involved intracranial surgery or device implantation.
8. Any other active implanted device.
9. Any previous brain surgery that would interfere with the placement of the leads or the functioning of the device.
10. A history of neurostimulation intolerance in any area of the body.
11. A condition requiring or likely to require the use of magnetic resonance imaging (MRI) or diathermy.
12. Currently on any anticoagulant medications that can not be discontinued during perioperative period.
13. Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, including any terminal illness with survival <12 months.
14. Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days. Any other trial participation should be approved by the Principal Investigators.
15. A female that is breastfeeding or of child bearing potential with a positive urine pregnancy test or not using adequate contraception.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Timmermann, M.D., Principal Investigator — Universitätsklinikum Köln; François Alesch, M.D., Principal Investigator — Allgemeines Krankenhaus AKH, Vienna, Austria
Locations (7):
- Allgemeines Krankenhaus AKH, Vienna, Austria
- CHU de Rennes-Pontchaillou, Rennes, France
- Uniklinik Köln, Cologne, Germany
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy
- Hospital Central de Asturias, Oviedo, Spain
- United Kingdom (2):
  - Frenchay Hospital, Bristol
  - Southmead Hospital Bristol, Bristol

REFERENCES:
- [Derived] Timmermann L, Jain R, Chen L, Maarouf M, Barbe MT, Allert N, Brucke T, Kaiser I, Beirer S, Sejio F, Suarez E, Lozano B, Haegelen C, Verin M, Porta M, Servello D, Gill S, Whone A, Van Dyck N, Alesch F. Multiple-source current steering in subthalamic nucleus deep brain stimulation for Parkinson's disease (the VANTAGE study): a non-randomised, prospective, multicentre, open-label study. Lancet Neurol. 2015 Jul;14(7):693-701. doi: 10.1016/S1474-4422(15)00087-3. Epub 2015 May 28. PMID 26027940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited at 6 European centers for the study
Groups:
- Deep Brain Stimulation: All enrolled subjects who met study eligiblity recieved Vercise DBS system as part of the study.
Period: Overall Study
Arm/Group | Deep Brain Stimulation
Started | 53
Completed | 39
Not Completed | 14
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 2
Not completed — not disclosed | 2
Not completed — Death | 1
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Population: 40 enrolled subjects who met study eligibility were implanted with the Vercise DBS system.
Groups:
- Deep Brain Stimulation: Vercise (TM) Rechargeable Deep Brain Stimulation System
  Deep Brain Stimulation: Rechargeable Deep Brain Stimulation System
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 40
Age, Customized [Number; unit: participants]
  <=60 years | 19
  61-70 years | 18
  >70 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 27
Region of Enrollment [Number; unit: participants]
  France | 1
  Spain | 11
  Austria | 12
  Germany | 9
  United Kingdom | 6
  Italy | 1

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change in UPDRS III Score From Baseline Meds Off to 12 and 52 Weeks Post First Lead Implantation Stim on/Meds Off.
Description: Unified Parkinson's Disease Rating Scale Part III (UPDRS III) is the motor sub-section of the Unified Parkinson's Disease Rating scale designed to evaluate overall motor disability, including the classic symptoms of Parkinson's Disease. This section has 14 items.
  Each item is scored on a scale from 0 (normal) to 4 (severe, marked, or unable), with the total possible score for the 14 items, including separate questions regarding symptoms present axially and in appendages, ranging from 0 to 108 with lower scores representing better results.
Time Frame: 12 and 52 weeks post first lead implantation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 40
units on a scale
  Mean Change from Baseline to Week 12 | -22.3 (8.05)
  Mean Change from Baseline to Week 52 | -23.7 (8.83)

2. Secondary Outcome: Mean Change in UPDRS II Score From Baseline Meds Off to 12, 26 and 52 Weeks Post First Lead Implantation Stim on/Meds Off.
Description: Unified Parkinson's Disease Rating Scale Part II (UPDRS II) is a sub-section of the Unified Parkinson's Disease Rating scale designed to evaluate Activities of Daily Living. This section contains 13 items.
  Each item is scored on a scale from 0 (normal) to 4 (disabled), with the total score for the 13 items ranging from 0 to 52.
Time Frame: 12, 26 and 52 weeks post first lead implantation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 40
units on a scale
  Change from Baseline to 12 weeks | -10.5 (7.76)
  Change from Baseline to 26 weeks | -11.8 (5.96)
  Change from Baseline to 52 weeks | -10.1 (8.55)

3. Secondary Outcome: Mean Change in Antiparkinsonian Medication Use in Mgs (Levodopa or Equivalents) From Baseline to 12, 26 and 52 Weeks Post First Lead Implantation
Description: All parkinsonian medications will be converted to Levodopa dose equivalents (LED) and baseline dose will be compared with dose taken at 12, 26 and 52 weeks post implantation
Time Frame: 12, 26 and 52 weeks post first lead implantation
Population: 40 completed Baseline, 35 completed Week12, 39 completed Week 26 and 38 completed Week 52
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 40
mg
  Change from Baseline to 12 weeks | -683.126 (537.91)
  Change from Baseline to 26 Weeks | -740 (603.6)
  Change from Baseline to 52 weeks | -816 (571.4)

4. Secondary Outcome: Mean Change in the Number of Waking Hours Per Day With Good Symptom Control and no Troublesome Dyskinesia From Baseline to 12, 26 and 52 Weeks Post First Lead Implantation.
Description: Subjects will complete a 3-day motor diary prior to study visits. At one-hour increments (during waking hours), patients will record "on", "on with troublesome dyskinesia", "off", and "asleep" times for three consecutive days.
Time Frame: 12, 26 and 52 weeks post first lead implantation
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 40
hours/day
  Change from Baseline to 12 weeks in ON time | 3.1 (7.3)
  Change from Baseline to 26 weeks in ON time | 3 (6.31)
  Change from Baseline to 52 weeks in ON time | 3.5 (6.58)

5. Secondary Outcome: Mean Percent Change in Quality of Life Scale Scores: Parkinson's Disease Questionnaire (PDQ-39) From Baseline Meds on to 12, 26 and 52 Weeks Post First Lead Implantation Stim on/Meds on.
Description: The Parkinson's Disease Questionnaire (PDQ-39) is a 39-item questionnaire designed to measure the specific impact of PD on quality of life. The questions measure the impact on health-related quality of life along 8 dimensions:
  * mobility
  * activities of daily living
  * emotional well-being
  * stigma
  * social support
  * cognitions
  * communication
  * bodily discomfort. Dimension scores range from 0 to 100, with 0 representing perfect health for the measure and 100 representing worst health for the measure.
Time Frame: 12, 26 and 52 weeks post first lead implantation
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 40
percentage change
  Percent Change from Baseline to 12 Weeks | -38 (41.2)
  Percent Change from Baseline to 26 Weeks | -29 (39)
  Percent Change from Baseline to 52 Weeks | -34.5 (45.6)

6. Secondary Outcome: Mean Percent Change in Quality of Life Scale Scores: Modified Schwab and England (SE) Scores From Baseline Meds on to 12, 26 and 52 Weeks Post First Lead Implantation Stim on/Meds on
Description: The purpose of the Schwab and England (SE) (13) single-item scale is to quantify a PD patients' ability to perform activities of daily living. The single item is based on a percentage rating with scores in 10% increments. Scores range from 0% (completely bed-ridden) to 100% (completely independent).
Time Frame: 12, 26 and 52 weeks post first lead implantation
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 40
percentage change
  Percent Change from baseline to 12 weeks | 9 (21)
  Percent Change from baseline to 26 weeks | 12 (26.2)
  Percent Change from Baseline to 52 weeks | 12.5 (23.4)

7. Primary Outcome: Mean Change in UPDRS III Score From Baseline in the Meds Off Condition (no Medications) to 26 Weeks Post First Lead Implantation in the Stim on/Meds Off Condition (Stimulation on and no Medications).
Description: as for outcome 1
Time Frame: 26 weeks post first lead implantation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 40
units on a scale | -23.8 (10.59)

8. Secondary Outcome: Percentage of Participants With Improved, No Change or Worsened Global Impression of Change (GIC) as Compared to Baseline, Evaluated by the Neurologist.
Description: Global Impression of Change (GIC) is a comparison to baseline and will be evaluated by rating the global impression of change using a seven-point scale: ("very much improved" to "marked worsening"). This assessment was completed by the neurologist.
Time Frame: 52 weeks post first lead implantation
Measure: Number; unit: percentage of participants
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 40
percentage of participants
  Percent Improved at 52 weeks | 97.4
  Percent with no change at 52 weeks | 0
  Percent worsened at 52 weeks | 2.6

ADVERSE EVENTS:
Arm/Group | Deep Brain Stimulation
Serious Adverse Events (participants affected / at risk) | 10/40
Other Adverse Events (participants affected / at risk) | 37/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Brain Stimulation (N=40)
Influenza (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Device migration (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Akinesia (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Brain Stimulation (N=40)
Fall (Injury, poisoning and procedural complications) | 9 (10)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 2 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 3 (3)
Dystonia (Nervous system disorders) | 2 (3)
Paraesthesia (Nervous system disorders) | 2 (2)
Parkinson's disease (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Cerebral microangiopathy (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Movement disorder (Nervous system disorders) | 1 (1)
Nerve root lesion (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 6 (6)
Apathy (Psychiatric disorders) | 3 (3)
Anger (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Impulse-control disorder (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Rapid eye movements sleep abnormal (Psychiatric disorders) | 1 (1)
Urinary tract infection (Reproductive system and breast disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (2)
Incision site infection (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (2)
Adverse drug reaction (General disorders) | 1 (1)
Axillary pain (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1)
Implant site haematoma (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Laboratory test abnormal (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No